CLINICAL TRIAL: NCT02039999
Title: An Investigation Into the Mechanism of Inhalation Cough Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ACADMED240913
Record Dates: First submitted 2013-12-16; First posted 2014-01-20 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Cough
Keywords: chronic; cough; challenge; ATP; hypersensitivity; TRPA1
MeSH Terms: conditions — Cough; Bronchiolitis Obliterans Syndrome; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chronic cough (Experimental): Cough challenges to be administered include:
  Nebulised citric acid in serial dilutions Nebulised ATP solution in serial dilutions Nebulised TRPA1 agonist solution in serial dilutions
  Interventions: Other: Nebulised citric acid in serial dilutions; Other: Nebulised ATP solution in serial dilutions; Other: Nebulised TRPA1 agonist solution in serial dilutions
- Normal volunteer (Active Comparator): Cough challenges to be administered include:
  Nebulised citric acid in serial dilutions Nebulised ATP solution in serial dilutions Nebulised TRPA1 agonist solution in serial dilutions
  Interventions: Other: Nebulised citric acid in serial dilutions; Other: Nebulised ATP solution in serial dilutions; Other: Nebulised TRPA1 agonist solution in serial dilutions

INTERVENTIONS:
Other: Nebulised citric acid in serial dilutions — Citric acid will be delivered in serial dilutions as per the clinical trials unit standard operating procedure for cough challenge using KoKo Digidoser, based on ERS guidelines. Challenge will be repeated until C5 (5 coughs in 30 seconds following challenge) is elicited.
Other: Nebulised ATP solution in serial dilutions — ATP solution will be delivered in serial dilutions as per the clinical trials unit standard operating procedure for cough challenge using KoKo Digidoser, based on ERS guidelines. Challenge will be repeated until C5 (5 coughs in 30 seconds following challenge) is elicited.
Other: Nebulised TRPA1 agonist solution in serial dilutions — TRPA1 agonist will be delivered in serial dilutions as per the clinical trials unit standard operating procedure for cough challenge using KoKo Digidoser, based on ERS guidelines. Challenge will be repeated until C5 (5 coughs in 30 seconds following challenge) is elicited.

SUMMARY:
Despite its commonplace use in respiratory medicine the mechanism whereby inhalation challenge with a variety of mild acid aerosols produces a dose related and predictable cough is unknown. In this proposal the investigators wish to use established cough challenge methodology to explore the mechanism of action of agents provoking cough both in health and disease.

The hypotheses to be tested include:

* Intracellular changes in pH, rather than extracellular changes, are key in the activation of TRP receptors, the main sensor for provoking cough.
* ATP acting through P2X channels is the mechanism of increased nerve excitability underlying cough hypersensitivity.

DETAILED DESCRIPTION:
The investigators have previously demonstrated that mild acids, such as citric, tartaric or phosphoric acid produce a highly reliable cough challenge and that the sensitivity of these are complex individual acids correlates within the population studied inferring a common mechanism of action.In contrast there is no correlation with the other common cough challenge methodology, capsaicin inferring that there are at least two different mechanisms for producing cough with aerosols in man.

Over the past 10 years it has been established that capsaicin works by a specific irritant receptor known as the TRPV1. A second receptor, TRPA1 has been recently discovered and we were the first group to demonstrate that inhalation of agonists of this receptor in the form of the extract of cinnamon (cinnamaldehyde) produces cough in man . TRPA1 is a very attractive candidate for the main cough receptor since it is activated by many common irritants, such as smoke, perfumes and other strong smells known to provoke coughing in patients.

The investigators have cloned the human TRP receptors and expressed them in cell lines. This in vitro work has allowed us to investigate the molecular action of the TRP receptors. Recently, the investigators and others have shown that weak acids can activate TRPA1, not as previously thought by stimulating the external surface of the cells but by altering the intracellular pH. This would explain why weak and not strong acids are better at producing cough, since weaker acids (technically those with a higher pKa) exist in solution in a form which is able to cross the cell membrane and render a change in the intracellular pH, which in turn activates TRPA1 from inside the cell.

In the first study the investigators wish to the simply alter the pH of the nebulised solution provoking cough by altering the balance of the salts in the solution, and then carry out standard cough challenge protocols.

In a second study the investigators wish to examine the effect of a number of known agonists of TRPA1 which are commonly used in the perfumes and foodstuffs in order to understand the rank order of potency of these compounds as tussive agents. This can then be compared to the rank order of potency of the same compounds in causing intracellular pH change in in vitro cell culture systems, in order to test the strength of the hypothesis over a variety of different agonists.

Finally, recent work has shown that blockade of a neuronal ion channel known as P2X3 can dramatically reduce cough. P2X3 responds to the substance adenosine triphosphate (ATP), which has previously been used as a cough challenge solution in man. If the hypothesis that the cough hypersensitivity seen in patients is due to activation of P2X3 is correct then patients will cough at much lower doses of ATP than normal volunteers. We wish to assess the value of ATP, and the related substance AMP and adenosine in a cough challenge protocol. Studying the cough produced by these naturally occurring compounds may allow us to distinguish patients with cough hypersensitivity from those with cough due to other causes, and also lead to a methodology important in future drug development

The greater understanding of the cough reflex which these studies would yield would have important clinical applications pointing the way to novel therapeutic avenues, as well as enhancing our fundamental understanding of the genesis of cough.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be required to demonstrate significant cough symptoms by a score greater than 20/70 on the Hull Airways Reflux Questionnaire.
* All patients must be current non-smokers.
* Patients must be on stable medication for at least one month.
* Patients must be able to attend the trials unit on at least 3 occasions.
* Patients must have normal lung function patients must be able to give informed consent

Exclusion Criteria:

* Subjects who are pregnant, or have pacemakers in situ are excluded from this study.
* Those with a serious comorbid conditions such as cancer, severe COPD, or heart failure will be excluded.
* Those who are non-English speakers and special groups (i.e. mentally ill, children under 16 years of age, and those suffering from dementia) will be excluded.
* No test will be performed on any subject during an acute worsening of asthma or upper airway infection. If the subject has had an upper airway infection in the last three weeks they will be offered another appointment.
* If the subject has taken any over the counter (OTC) cough mixture within the last twelve hours: If the subject is willing to come back another time for challenge testing, another appointment should be made.
* If the subject has had any food or drink products containing caffeine or menthol within the last hour. If the subject is unwilling to wait for 1 hour before starting the test, the subject should return another time. If the subject is unwilling to return another time, testing should proceed and the medication used recorded.
* If the participant is currently involved in research, or within 3 months of participation in any type of research, they will be excluded from this study.

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Difference in mean C5 (concentration of inhaled substance required to elicit 5 coughs) (ATP) and total cough (citric acid) between the chronic cough arm and the normal volunteer arm. | Coughs will be measured in a 30 second period following the inhalation of each challenge substance.
  Following inhalation of challenge substance, subject will be monitored for 30 seconds and number of coughs recorded. Concentration of challenge substance will increase until subject coughs at least 5 times following challenge. This will be recorded as the C5 value for each subject. The mean C5 value will be compared between the chronic cough arm and the normal volunteer arm. This will be reported as whether or not there is a statistical difference between the mean C5 for the chronic cough group and the normal volunteer group.

CONTACTS AND LOCATIONS:
Overall Officials: Alyn H Morice, MD, FRCP, Principal Investigator — National Health Service, United Kingdom
Locations (1):
- Hull Clinical Trials Unit, Respiratory academic department, Cottingham, East Yorkshire, United Kingdom

REFERENCES:
- [Background] Fowles HE, Rowland T, Wright C, Morice A. Tussive challenge with ATP and AMP: does it reveal cough hypersensitivity? Eur Respir J. 2017 Feb 8;49(2):1601452. doi: 10.1183/13993003.01452-2016. Print 2017 Feb. PMID 28179439
- See also: Publication Link — https://erj.ersjournals.com/content/49/2/1601452